CLINICAL TRIAL: NCT02858466
Title: Structural and Functional Brain Reorganization in Neuropathic Pain: Basal State of Local Cerebral Blood Flow and Functional Connectivity
Acronym: CONNECT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: failure to recruit
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1308144; 2013-A01440-45 (Other: ANSM)
Record Dates: First submitted 2016-07-25; First posted 2016-08-08 (Estimated); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- peripheric nervous lesion (Experimental): MRI scan
  Interventions: Radiation: MRI scan
- medullar or encephalic lesion (Experimental): MRI scan
  Interventions: Radiation: MRI scan
- control group (Other): MRI scan
  Interventions: Radiation: MRI scan

INTERVENTIONS:
Radiation: MRI scan

SUMMARY:
Neuropathic pain is a medical condition involving allodynia (painful perceptions in response to stimuli that normally are not) and spontaneous pain (occurring at rest, without stimulation).

This pain is secondary to nervous system injury affecting the sensory system. The lesion is either at the nerve endings of the spinal cord or brain.

It induces a loss of sensitivity and likely reorganization of brain activity that are causing pain and which are the subject of this study.

Previous studies in functional neuroimaging has focused on brain areas activated during allodynic stimuli compared to non-painful stimuli. The abnormalities have been reported, but it was not possible to conclude formally. The authors failed to assess the part of the effect of the loss of sensory afferents (deafferentation) and the basal brain function.

Indeed, the operation without any sensory stimulation is not known yet is the initial level of activity which is the benchmark for studying brain function during stimulation. The objective of this study is to understand what are the cortical systems of allodynic dysfunctional in patients compared with controls at baseline.

ELIGIBILITY:
Inclusion Criteria for patients :

* major
* with nervous pain : chronic or peripheric
* treatment not stable opioid since one week
* signed consent

Inclusion Criteria for witnesses :

* major
* without chronic pain
* signed consent

Exclusion Criteria for 2 groups :

* severe psychiatric history
* presence of an active nervous lesion
* subject with morphine treatment
* contraindication to MRI scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-03-25 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
cerebral blood flow | at baseline
  quantified with MRI scan

SECONDARY OUTCOMES:
rate of grey matter | at baseline
  difference between groups
structure of the networks | at baseline
  Determine if structure of the networks is different between patients and controls.
  Measured with MRI scan.
connection of the networks | at baseline
  Determine if connection of the networks is different between patients and controls.
  Measured with MRI scan.
cortical loss | at baseline
  Assess the cortical loss of the patient group compared to controls. Measured with MRI scan.

CONTACTS AND LOCATIONS:
Overall Officials: Roland PEYRON, MD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No